CLINICAL TRIAL: NCT06274281
Title: Implementing a Digital Telerehabilitation Protocol and Non-motor Outcomes, and Quality of Life in Patients With Functional Motor Disorders: a Feasibility 2-arm Parallel Randomized Controlled Clinical Trial
Brief Title: Digital Telerehabilitation in Functional Motor Disorders
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Marialuisa Gandolfi, Full Professor, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TOMs_FMD
Record Dates: First submitted 2024-01-19; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Functional Movement Disorder
Keywords: Gait; Wearable devices; Digital telerehabilitation
MeSH Terms: conditions — Conversion Disorder

STUDY DESIGN:
Intervention Model Description: This is an experimental single-blind randomized-controlled trial (RCT) with 2-parallel arms comparing the effects between the experimental group (EG) and control group (CG). After screening, a simple randomization list will be generated by a physician using an automated randomization system (alloca-tion ratio 1:1) to assign eligible patients to either the EG or the CG. Group allocation will be kept concealed.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be blinded to the type of intervention performed by the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group Training (Experimental): After the intensive 5-days rehabilitation treatment (2 hours/day, 5 days/week, for 1 week), the EG pa-tients will be encouraged to perform the self-management plan at home with the same duration and in-tensity as the CG (1 hour/session, 3 sessions/week, 12 weeks) through a Digital Telemedicine platform (Phoema GPI Platform, GPI Spa, Trento, Italy). The platform will be implemented with wearable digital devices Axivity AX3, 3-axis Logging Accel-erometer to gather objective and subjective information on the patient's motor activity. At discharge (T1), each patient in the experimental group will receive 2 wearable sensors (Axivity AX3,) for moni-toring of movement data (i.e., activity level, number of steps, distance travelled). The data will be transmitted periodically to the research center and processed. The subjective assessment of the patient's motor activity will be collected by clinical diaries focusing on gait and activity level.
  Interventions: Device: Digital Telerehabilitation
- Control Group Training (Active Comparator): After the intensive 5-days rehabilitation treatment (2 hours/day, 5 days/week, for 1 week), the CG patients will be encouraged to perform the self-management plan at home with the same duration and intensity as the EG (1 hour/session, 3 sessions/week, 12 weeks) without a Digital Telemedicine platform and wearable devices use.
  Interventions: Other: Usual care

INTERVENTIONS:
Device: Digital Telerehabilitation — The 5-day rehabilitation program will consist of exercises to re-establish standard movement patterns within a multidisciplinary etiological framework, according to a validated rehabilitation protocol for FMDs. Treatment will be tailored to the needs of each patient, following general treatment principles in physiotherapy for FMDs.
  Telemedicine sessions: the patient will perform specific exercises under the supervision of a qualified physiotherapist to provide feedback on the execution and adapt the treatment according to clinical changes/improvements.
  Wearable devices: each patient in the experimental group will receive 2 wearable sensors (Axivity AX3,) for monitoring of movement data (i.e., activity level, number of steps, distance travelled) during daylife activities and rehabilitation sessions. The subjective assessment of the patient's motor activity will be collected by clinical diaries focusing on gait and activity level.
  Arms: Experimental Group Training
Other: Usual care — The 5-day rehabilitation program will be the same as the telemedicine group. A self-management paper log will be given to the patient at the end of the 5-day rehabilitation program. It will include goals, activity plans, and strategies to be used for retraining movements and redirecting attention. Videos stored on the patients' digital device (i.e., tablet, mobile) will include exercises demonstration and execution and strategies to retrain movements. Patients will be encouraged to perform the self-management plan at home on their own (or with their caregivers' help) which will be reported in a paper log and video recorded. The subjective assessment of the patient's motor activity will be collected by clinical diaries focusing on gait and activity level.
  Arms: Control Group Training

SUMMARY:
Functional motor disorders (FMDs) are a broad spectrum of functional neurological disorders, including abnormal gait/balance disorders. Patients experience high degrees of disability and distress, equivalent to those suffering from degenerative neurological diseases. Rehabilitation is essential in their management. However, the current systems of rehabilitation delivery face two main challenges. Patients are not receiving the amount and kind of evidence-based rehabilitation they need due to the lack of rehabilitation professionals and experts in the field. The rehabilitation setting is not adequate for the long-term management and monitoring of these patients. Digital medicine is a new field that means "using digital tools to upgrade the practice of medicine to one that is high-definition and far more individualized." It can upgrade rehabilitation practice, addressing the existing critical components towards marked efficiency and productivity. Digital telerehabilitation will increase the accessibility to personalized rehabilitation by expert professionals placing tools to monitor the patient's health by themselves.

The increasing development and availability of portable and wearable technologies are rapidly expanding the field of technology-based objective measures (TOMs) in neurological disorders. However, substantial challenges remain in (1) recognizing TOMs relevant to patients and clinicians to provide accurate, objective, and real-time assessment of gait and activity in a real-world setting and (2) their integration into telerehabilitation systems towards a digital rehabilitation transition.

This feasibility study provides preliminary data on the integration of a real-time gait and activity analysis by wearable devices in the real world with a digital platform to improve the diagnosis, monitoring, and rehabilitation of patients with FMDs.

DETAILED DESCRIPTION:
Functional movement disorders (FMDs) are part of a wide spectrum of functional neurological disorders characterized by abnormal movements (gait, dystonia, and tremor), which are clinical incongruent with movement disorders caused by neurological disease and are significantly altered by distraction or nonphysiologically manoeuvres. FMDs have an incidence ranging from 4 to 12 per 100.000 population per year and high prevalence (15-20%) in patients accessing neurological clinics. They are a high disabling condition characterized by long-term disability, poor quality of life and economic impact on health and social care systems. Indeed, these patients experience disability and distress equivalent to those suffering from degenerative neurological disease, such as Parkinson's Disease. Despite this, FMDs have been widely misunderstood, receiving little public and academic attention.

Diagnostic clinical criteria for FMDs are based on positive signs that support certain integrity of the pathway from an anatomical and physiological perspective: specific maneuvers can make apparent the function that seems to be lost or impaired. Despite the clinical burden, the exact pathophysiological mechanisms underlying FMDs have not been elucidated and so FMDs' management remain largely unknown. The hallmarks of FMDs patients distinguishing them from those with organic movement disorders is that their movements have features usually associated with voluntary movement. Still, patients report them as involuntary and not under their control. Why movements that appear voluntary because altered by distraction are experienced as involuntary (or outside the patient's control) is a matter of debate.

In addition to motor complaints, non-motor symptoms (NMSs) such as fatigue, pain, anxiety, depression have been increasingly recognized as important contributors producing levels of disability over and above those caused by the abnormal movement. Within this perspective should be considered the rehabilitation of patients with FMDs, to reduce disability and improve Health-related Quality of Life (QoL) in the context of a multidisciplinary team. To do that, there are limits that must be overcome: rehabilitation approaches are few and limited because of empirical approaches mainly referring to clinical practice without following evidence-based consensus recommendations, most existing studies are uncontrolled case series or crossover studies and innovations to improve access to specialist rehabilitation treatment by qualified professionals (i.e., tele/remote health an wearable technology) and to monitor patients in the long-term have been seldom explored in patients with FMDs.

Digital medicine, a new field based on "using digital tools to upgrade the practice of medicine to one that is high-definition and far more individualized", led the introduction of a new path for generating a new form of healthcare through the medical data acquisition by the individual, in real time, in a real-world environment, enabling site-less, digital clinical trials where suitable participants are identified, consented, and enrolled remotely. The next phase of this will greatly impact clinicians across disciplines including rehabilitation. In fact, in the last few years, telerehabilitation (a telemedicine subfield consisting of a system to control rehabilitation at a distance) has been progressively developed allowing to overcome the barrier of distance and time (mainly in communities far from urban centers), to cut down the cost and labor of accessing healthcare, and to provide access to patients having temporary and permanent disabilities for accurate diagnosis and rehabilitation prescription and delivery.

Digital telerehabilitation combined the advantages of telerehabilitation with the possibility to use digital tools (i.e., wearable sensors, digital platform) in monitoring functions and activities in real-time and in the real-world environment. Digital Telemedicine platforms offer new opportunities for diagnosis, monitoring, treatment, and management of diseases allowing the acquisition, transmission, and storage of clinical information through electronic devices and communication technologies to provide and support remote health care, including rehabilitation. The use of digital technologies applied to rehabilitation through telemedicine systems (telerehabilitation) represents one of the main fronts of development in neurological rehabilitation as it offers the potential to extend specific rehabilitation paths from the hospital phase to the home phase allowing, thanks to the involvement of highly qualified personnel, better management of diseases and their clinical, social and economic outcomes.

The increasing development and availability of portable and wearable technologies are rapidly expanding the field of technology-based objective measures (TOMs) in neurological disorders. However, substantial challenges remain in (1) recognizing TOMs relevant to patients and clinicians to provide accurate, objective, and real-time assessment of gait and activity in a real-world setting and (2) their integration into telerehabilitation systems towards a digital rehabilitation transition. It is crucial in FMDs because of the clinical complexity of patients who require highly qualified personnel, adapting rehabilitation programs over time according to the patients' improvements, and long-term monitoring without impacting health care costs. Besides the pandemic caused by the SARS-CoV-2 virus, which has prevented patients from accessing rehabilitation in hospital settings, the restricted presence of qualified centers for the rehabilitation of patients with FMDs emphasizes the need to create specific digital telerehabilitation pathways by qualified staff that can reach patients who would not have access to such rehabilitative treatment. However, pilot studies for phase III trials - which are comparative randomized trials designed to provide preliminary evidence on the clinical efficacy of a drug or intervention (also commonly known as "feasibility" studies), must be designed to assess the safety of treatment or interventions; to assess recruitment potential; to assess the feasibility of international collaboration or coordination for multicenter trials; to increase clinical experience with the study medication or intervention for the phase III trials . They are the best way to assess feasibility of a large, expensive full-scale study, and in fact are an almost essential pre-requisite.

The primary aim of the study is to implement and assess the feasibility of the steps that need to take place as part of the main confirmatory study on comparing the effects of a digital telerehabilitation program including TOMs on motor symptoms severity and duration in patients with FMDs. The secondary aim is then to compare the training effects on non-motor symptoms (pain, fatigue, anxiety and depression), the self-perception of clinical change and Health-Related Quality of Life, and health care costs.

ELIGIBILITY:
Inclusion Criteria:

* a clinically definite diagnosis of FMDs based on Gupta and Lang diagnostic criteria with the presence of distractibility maneuvers and a demonstration of positive signs
* the presence of 1 (isolated FMDs) or more clinical motor symptoms (combined FMDs), including weakness, tremor, jerks, dystonia, gait disorders, and parkinsonism
* acceptance of the diagnosis on the balance of probability
* severity and duration of motor impairment ≥1 scored with the Simplified Functional Movement Disorders Rating Scale (SFMDRS)
* acceptable level of digital skills.

Exclusion Criteria:

* Prominent dissociative seizures
* Mini-Mental State Examination <23/30
* Patients who continue to express some doubt over the diagnosis.
* prominent cognitive and physical impairment that preclude signing the informed consent for participation in the study.
* Unable or refuse to attend the consecutive 5-day rehabilitation treatment. Patients will give their written informed consent after being informed about the experimental nature of the study. According to the Helsinki Declaration, the study will be carried out, approved by the Local Ethics Committee, and registered at the clinical trial.
* Particularly vulnerable population. The following cannot be included in the study: pregnant women, patients in an emergency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
number of patients who accept/refuse the treatment, physiotherapy compliance and falls or event near falling occurred during rehabilitation | before the intensive 5-day rehabilitation program (T0), the day after the intensive 5-day rehabilitation program (T1), after 12 weeks (at the end of the self-management plan, T2), and 24 weeks (follow-up, T3)
  recruitment rate, acceptability of the intervention in terms of number of dropouts before the end of treatment, and safety in terms of reported adverse events during the treatment.
Budget issues related to TOMs | before the intensive 5-day rehabilitation program (T0), the day after the intensive 5-day rehabilitation program (T1), after 12 weeks (at the end of the self-management plan, T2), and 24 weeks (follow-up, T3)
  Budget issues in the use of TOMs during the EG intervention
Time spent to train patients | before the intensive 5-day rehabilitation program (T0), the day after the intensive 5-day rehabilitation program (T1), after 12 weeks (at the end of the self-management plan, T2), and 24 weeks (follow-up, T3)
  Time to train the patient in using the TOMs

SECONDARY OUTCOMES:
Change in the Simplified Functional Movement Disorders Rating Scale (S-FMDRS) score | before the intensive 5-day rehabilitation program (T0), the day after the intensive 5-day rehabilitation program (T1), after 12 weeks (at the end of the self-management plan, T2), and 24 weeks (follow-up, T3)
  Objective-rated validated scale to rate the duration and severity of functional motor symptoms (range: 0-54; higher = worse).
Multidimensional Fatigue Inventory Scale (MFI-20) score | before the intensive 5-day rehabilitation program (T0), the day after the intensive 5-day rehabilitation program (T1), after 12 weeks (at the end of the self-management plan, T2), and 24 weeks (follow-up, T3)
  It evaluates fatigue differentiating general, physical, reduced-activity, reduced-motivation, and mental fatigue (subscale range: 4-20; higher = worse).
Change in the Brief Pain Inventory (BPI) score | before the intensive 5-day rehabilitation program (T0), the day after the intensive 5-day rehabilitation program (T1), after 12 weeks (at the end of the self-management plan, T2), and 24 weeks (follow-up, T3)
  It evaluates pain intensity (range: 0-40; higher = worse) and interference (range: 0-70; higher = worse).
Change in the Beck Depression Inventory (BDI-II) score | before the intensive 5-day rehabilitation program (T0), the day after the intensive 5-day rehabilitation program (T1), after 12 weeks (at the end of the self-management plan, T2), and 24 weeks (follow-up, T3)
  It evaluates depression (range: 0-63; higher = worse).
Change in the Beck Anxiety Inventory (BAI) score | before the intensive 5-day rehabilitation program (T0), the day after the intensive 5-day rehabilitation program (T1), after 12 weeks (at the end of the self-management plan, T2), and 24 weeks (follow-up, T3)
  It evaluates anxiety (range: 0-63; higher = worse).
Change in the 12-item Short-Form Health Survey (SF-12) score | before the intensive 5-day rehabilitation program (T0), after 12 weeks (at the end of the self-management plan, T2), and 24 weeks (follow-up, T3)
  The health-Related QoL will be evaluated by the Mental Health and Physical functioning of the 12-item Short-Form Health Survey (SF-12) (range: 0-100; higher = better)
The EuroQol-5D (EQ-5D) | before the intensive 5-day rehabilitation program (T0), after 12 weeks (at the end of the self-management plan, T2), and 24 weeks (follow-up, T3)
  It evaluates generic quality of life. The scale ranges from 100 ('the best imaginable health state' or 'the best health state you can imagine') to 0 ('the worst imaginable health state' or 'the worst health you can imagine').
iMTA Productivity Cost Questionnaire | before the intensive 5-day rehabilitation program (T0), after 12 weeks (at the end of the self-management plan, T2), and 24 weeks (follow-up, T3)
  It is a Standardized Instrument for Measuring and Valuing Health-Related Productivity Losses. Index score can vary from 0 to 21, with higher scores indicating better quality of life.
Change in the Clinical Global Impression (CGI) score | the day after the intensive 5-day rehabilitation program (T1), after 12 weeks (at the end of the self-management plan, T2), and 24 weeks (follow-up, T3
  Self-rated perception of change will be assessed with the 7-point Clinical Global Impression (CGI) scale with scores from 1 (very much improved) to 7 (very much worse).
Gait outcome: Gait speed | before the intensive 5-day rehabilitation program (T0), the day after the intensive 5-day rehabilitation program (T1), after 12 weeks (at the end of the self-management plan, T2), and 24 weeks (follow-up, T3)
  They will be evaluated at hospital with Axivity AX3. The outcome for gait will be gait speed (cm/s)
Gait outcome: Stride length | before the intensive 5-day rehabilitation program (T0), the day after the intensive 5-day rehabilitation program (T1), after 12 weeks (at the end of the self-management plan, T2), and 24 weeks (follow-up, T3)
  They will be evaluated at hospital with Axivity AX3. The outcome for gait will be stride length (cm).
Gait outcome: Cadence | before the intensive 5-day rehabilitation program (T0), the day after the intensive 5-day rehabilitation program (T1), after 12 weeks (at the end of the self-management plan, T2), and 24 weeks (follow-up, T3)
  They will be evaluated at hospital with Axivity AX3. The outcome for gait will be cadence (step/min)
Balance outcome: CoP trajectory | before the intensive 5-day rehabilitation program (T0), the day after the intensive 5-day rehabilitation program (T1), after 12 weeks (at the end of the self-management plan, T2), and 24 weeks (follow-up, T3)
  They will be evaluated at hospital stabilometric platform. The outcome for postural control will be the length of the centre of pressure (CoP) trajectory (mm) measured in the eyes open (integrating visual, proprioceptive, and vestibular contributions) and the eyes closed condition (proprioceptive contribution to and the visual dependency on postural control).
Balance outcomes: Sway area | before the intensive 5-day rehabilitation program (T0), the day after the intensive 5-day rehabilitation program (T1), after 12 weeks (at the end of the self-management plan, T2), and 24 weeks (follow-up, T3)
  They will be evaluated at hospital stabilometric platform. The outcome for postural control will be the sway area (mm2) measured in the eyes open (integrating visual, proprioceptive, and vestibular contributions) and the eyes closed condition (proprioceptive contribution to and the visual dependency on postural control).

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Department of Neurosciences, Biomedicine and Movement Sciences, University of Verona, Verona
  - USD Parkinson's Disease and Movement Disorders Unit, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carson A, Lehn A. Chapter 5 Epidemiology. Published online 2016. doi:10.1016/B978-0-12-801772- 2.00005-9
- [Background] Edwards MJ, Bhatia KP. Functional (psychogenic) movement disorders: merging mind and brain. Lancet Neurol. 2012 Mar;11(3):250-60. doi: 10.1016/S1474-4422(11)70310-6. PMID 22341033
- [Background] Barbey A, Aybek S. Functional movement disorders. Curr Opin Neurol. 2017 Aug;30(4):427-434. doi: 10.1097/WCO.0000000000000464. PMID 28590986
- [Background] Erro R, Brigo F, Trinka E, Turri G, Edwards MJ, Tinazzi M. Psychogenic nonepileptic seizures and movement disorders: A comparative review. Neurol Clin Pract. 2016 Apr;6(2):138-149. doi: 10.1212/CPJ.0000000000000235. PMID 27104066
- [Background] Popkirov S, Nicholson TR, Bloem BR, Cock HR, Derry CP, Duncan R, Dworetzky BA, Edwards MJ, Espay AJ, Hallett M, Lang AE, Leach JP, Lehn A, McGonigal A, Morgante F, Perez DL, Reuber M, Richardson MP, Smith P, Stamelou M, Tijssen MAJ, Tinazzi M, Carson AJ, Stone J. Hiding in Plain Sight: Functional Neurological Disorders in the News. J Neuropsychiatry Clin Neurosci. 2019 Fall;31(4):361-367. doi: 10.1176/appi.neuropsych.19010025. Epub 2019 May 23. PMID 31117907
- [Background] Espay AJ, Aybek S, Carson A, Edwards MJ, Goldstein LH, Hallett M, LaFaver K, LaFrance WC Jr, Lang AE, Nicholson T, Nielsen G, Reuber M, Voon V, Stone J, Morgante F. Current Concepts in Diagnosis and Treatment of Functional Neurological Disorders. JAMA Neurol. 2018 Sep 1;75(9):1132-1141. doi: 10.1001/jamaneurol.2018.1264. PMID 29868890
- [Background] Edwards MJ. Neurobiologic theories of functional neurologic disorders. Handb Clin Neurol. 2017;139:131-137. doi: 10.1016/B978-0-12-801772-2.00012-6. PMID 27719834
- [Background] Aybek S, Nicholson TR, O'Daly O, Zelaya F, Kanaan RA, David AS. Emotion-motion interactions in conversion disorder: an FMRI study. PLoS One. 2015 Apr 10;10(4):e0123273. doi: 10.1371/journal.pone.0123273. eCollection 2015. PMID 25859660
- [Background] Voon V, Cavanna AE, Coburn K, Sampson S, Reeve A, LaFrance WC Jr; (On behalf of the American Neuropsychiatric Association Committee for Research). Functional Neuroanatomy and Neurophysiology of Functional Neurological Disorders (Conversion Disorder). J Neuropsychiatry Clin Neurosci. 2016 Summer;28(3):168-90. doi: 10.1176/appi.neuropsych.14090217. Epub 2016 Feb 22. PMID 26900733
- [Background] Kilteni K, Bergstrom I, Slater M. Drumming in immersive virtual reality: the body shapes the way we play. IEEE Trans Vis Comput Graph. 2013 Apr;19(4):597-605. doi: 10.1109/TVCG.2013.29. PMID 23428444
- [Background] Yee, N., and Bailenson, J. The proteus effect: the effect of transformed self-representation on behavior. Hum. Commun. Res. 2007;33:271-290.
- [Background] Gupta A, Lang AE. Psychogenic movement disorders. Curr Opin Neurol. 2009 Aug;22(4):430-6. doi: 10.1097/WCO.0b013e32832dc169. PMID 19542886
- [Background] Haggard P, Chambon V. Sense of agency. Curr Biol. 2012 May 22;22(10):R390-2. doi: 10.1016/j.cub.2012.02.040. No abstract available. PMID 22625851
- [Background] Nielsen G, Ricciardi L, Meppelink AM, Holt K, Teodoro T, Edwards M. A Simplified Version of the Psychogenic Movement Disorders Rating Scale: The Simplified Functional Movement Disorders Rating Scale (S-FMDRS). Mov Disord Clin Pract. 2017 Mar 11;4(5):710-716. doi: 10.1002/mdc3.12475. eCollection 2017 Sep-Oct. PMID 30363505
- [Background] Plummer P, Eskes G. Measuring treatment effects on dual-task performance: a framework for research and clinical practice. Front Hum Neurosci. 2015 Apr 28;9:225. doi: 10.3389/fnhum.2015.00225. eCollection 2015. PMID 25972801
- [Background] Nielsen G, Buszewicz M, Stevenson F, Hunter R, Holt K, Dudziec M, Ricciardi L, Marsden J, Joyce E, Edwards MJ. Randomised feasibility study of physiotherapy for patients with functional motor symptoms. J Neurol Neurosurg Psychiatry. 2017 Jun;88(6):484-490. doi: 10.1136/jnnp-2016-314408. Epub 2016 Sep 30. PMID 27694498
- [Background] Gandolfi M, Riello M, Bellamoli V, Bombieri F, Geroin C, Di Vico IA, Tinazzi M. Motor and non-motor outcomes after a rehabilitation program for patients with Functional Motor Disorders: A prospective, observational cohort study. NeuroRehabilitation. 2021;48(3):305-314. doi: 10.3233/NRE-201617. PMID 33780378
- [Background] Nielsen G, Stone J, Edwards MJ. Physiotherapy for functional (psychogenic) motor symptoms: a systematic review. J Psychosom Res. 2013 Aug;75(2):93-102. doi: 10.1016/j.jpsychores.2013.05.006. Epub 2013 Jun 12. PMID 23915764
- [Background] Gandolfi M, Fiorio M, Geroin C, Prior M, De Marchi S, Amboni M, Smania N, Tinazzi M. Motor dual task with eyes closed improves postural control in patients with functional motor disorders: A posturographic study. Gait Posture. 2021 Jul;88:286-291. doi: 10.1016/j.gaitpost.2021.06.011. Epub 2021 Jun 11. PMID 34153806
- [Background] W.G. (1976). Clinical global impression scale. The ECDEU Assessment Manual for Psychopharmacology, Revised. US Department of Health, Education, and Welfare Publication (ADM), 76(338):218-222.
- [Background] Geroin C, Gandolfi M, Maddalena I, Smania N, Tinazzi M. Do Upper and Lower Camptocormias Affect Gait and Postural Control in Patients with Parkinson's Disease? An Observational Cross-Sectional Study. Parkinsons Dis. 2019 Jul 24;2019:9026890. doi: 10.1155/2019/9026890. eCollection 2019. PMID 31428306
- [Background] Marotta A, Bombieri F, Zampini M, Schena F, Dallocchio C, Fiorio M, Tinazzi M. The Moving Rubber Hand Illusion Reveals that Explicit Sense of Agency for Tapping Movements Is Preserved in Functional Movement Disorders. Front Hum Neurosci. 2017 Jun 6;11:291. doi: 10.3389/fnhum.2017.00291. eCollection 2017. PMID 28634447
- [Background] Tinazzi M, Geroin C, Erro R, Marcuzzo E, Cuoco S, Ceravolo R, Mazzucchi S, Pilotto A, Padovani A, Romito LM, Eleopra R, Zappia M, Nicoletti A, Dallocchio C, Arbasino C, Bono F, Pascarella A, Demartini B, Gambini O, Modugno N, Olivola E, Bonanni L, Antelmi E, Zanolin E, Albanese A, Ferrazzano G, de Micco R, Lopiano L, Calandra-Buonaura G, Petracca M, Esposito M, Pisani A, Manganotti P, Stocchi F, Coletti Moja M, Antonini A, Ercoli T, Morgante F. Functional motor disorders associated with other neurological diseases: Beyond the boundaries of "organic" neurology. Eur J Neurol. 2021 May;28(5):1752-1758. doi: 10.1111/ene.14674. Epub 2021 Jan 2. PMID 33300269
- [Background] Tinazzi M, Morgante F, Marcuzzo E, Erro R, Barone P, Ceravolo R, Mazzucchi S, Pilotto A, Padovani A, Romito LM, Eleopra R, Zappia M, Nicoletti A, Dallocchio C, Arbasino C, Bono F, Pascarella A, Demartini B, Gambini O, Modugno N, Olivola E, Di Stefano V, Albanese A, Ferrazzano G, Tessitore A, Zibetti M, Calandra-Buonaura G, Petracca M, Esposito M, Pisani A, Manganotti P, Stocchi F, Coletti Moja M, Antonini A, Defazio G, Geroin C. Clinical Correlates of Functional Motor Disorders: An Italian Multicenter Study. Mov Disord Clin Pract. 2020 Sep 22;7(8):920-929. doi: 10.1002/mdc3.13077. eCollection 2020 Nov. PMID 33163563
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-15: validity of a new measure for evaluating the severity of somatic symptoms. Psychosom Med. 2002 Mar-Apr;64(2):258-66. doi: 10.1097/00006842-200203000-00008. PMID 11914441
- [Background] Kizony, R., Katz, N., Rand, D., & Weiss, P. L. T. (2006, December). Short Feedback Questionnaire (SFQ) to enhance client-centered participation in virtual environments. In Cyberpsychology & Behavior (Vol. 9, No. 6, pp. 687-688).
- [Background] Perez DL, Edwards MJ, Nielsen G, Kozlowska K, Hallett M, LaFrance WC Jr. Decade of progress in motor functional neurological disorder: continuing the momentum. J Neurol Neurosurg Psychiatry. 2021 Mar 15:jnnp-2020-323953. doi: 10.1136/jnnp-2020-323953. Online ahead of print. PMID 33722822
- [Background] Crea S, D'Alonzo M, Vitiello N, Cipriani C. The rubber foot illusion. J Neuroeng Rehabil. 2015;12:77. Robert S. Kennedy , Norman E. Lane, et. al. Simulator Sickness Questionnaire: An Enhanced Method for Quantifying Simulator Sickness, The International Journal of Aviation Psychology, 1993;3:203-220.
- [Background] Demartini B, Bombieri F, Goeta D, Gambini O, Ricciardi L, Tinazzi M. A physical therapy programme for functional motor symptoms: A telemedicine pilot study. Parkinsonism Relat Disord. 2020 Jul;76:108-111. doi: 10.1016/j.parkreldis.2019.05.004. Epub 2019 May 3. PMID 31078400
- [Background] Lubetzky AV, Kary EE, Harel D, Hujsak B, Perlin K. Feasibility and reliability of a virtual reality oculus platform to measure sensory integration for postural control in young adults. Physiother Theory Pract. 2018 Dec;34(12):935-950. doi: 10.1080/09593985.2018.1431344. Epub 2018 Jan 24. PMID 29364733
- [Background] Cortes-Perez I, Nieto-Escamez FA, Obrero-Gaitan E. Immersive Virtual Reality in Stroke Patients as a New Approach for Reducing Postural Disabilities and Falls Risk: A Case Series. Brain Sci. 2020 May 15;10(5):296. doi: 10.3390/brainsci10050296. PMID 32429085
- [Background] Gandolfi M, Sandri A, Geroin C, Bombieri F, Riello M, Menaspa Z, Bonetto C, Smania N, Tinazzi M. Improvement in motor symptoms, physical fatigue, and self-rated change perception in functional motor disorders: a prospective cohort study of a 12-week telemedicine program. J Neurol. 2022 Nov;269(11):5940-5953. doi: 10.1007/s00415-022-11230-8. Epub 2022 Jul 9. PMID 35809125
- [Background] Buchholz I, Janssen MF, Kohlmann T, Feng YS. A Systematic Review of Studies Comparing the Measurement Properties of the Three-Level and Five-Level Versions of the EQ-5D. Pharmacoeconomics. 2018 Jun;36(6):645-661. doi: 10.1007/s40273-018-0642-5. PMID 29572719
- [Background] Thabane L, Ma J, Chu R, Cheng J, Ismaila A, Rios LP, Robson R, Thabane M, Giangregorio L, Goldsmith CH. A tutorial on pilot studies: the what, why and how. BMC Med Res Methodol. 2010 Jan 6;10:1. doi: 10.1186/1471-2288-10-1. PMID 20053272